CLINICAL TRIAL: NCT03175250
Title: Action Plans & Memory Consolidation: Reducing HIV Risk in Drug Users
Brief Title: Translation of Basic Research in Cognitive Science to HIV Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Claremont Graduate University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Alan Stacy, Professor, Claremont Graduate University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: 1R01DA033871 (NIH); 1R01DA033871 (NIH)
Record Dates: First submitted 2017-06-01; First posted 2017-06-05 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned at the individual level to one of three different conditions within each drug diversion class.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants were randomly assigned by computer algorithm to three different conditions, and the intervention took place over individually assigned computers with screens that were not observable by the care provider, investigator, or outcome assessor. The two control groups were designed to be "active," that is, designed to have some effects. Thus, there was no indication of which intervention might be more effective.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Health Education (Active Comparator): This condition included live health education followed by health education videos on HIV risks, testing, and condom use. The videos were presented over laptop.
  Interventions: Behavioral: Health Education
- Action Plan (Active Comparator): This condition included live health education followed by computerized procedures focusing on action plans for HIV testing and condom use and some of the same health education videos in the Health Education condition.
  Interventions: Behavioral: Action Plan
- Memory Practice (Experimental): This condition included live health education followed by computerized action plan procedures (as in the Action Plan condition), followed by several memory practice procedures also delivered over laptop. The memory practice procedures were designed to help participants more readily retrieve and use action plans in critical situations.
  Interventions: Behavioral: Memory Practice

INTERVENTIONS:
Behavioral: Health Education — Videos (AIDSvideos.org) were presented on individually-assigned laptops and covered HIV risk, condom use, safe sex, and infection testing
  Arms: Health Education
Behavioral: Action Plan — Participants selected situations for condom use and screening for HIV and hepatitis on individually-assigned laptops. They linked these situations to preventive behaviors regarding screening and condom use.
  Arms: Action Plan
Behavioral: Memory Practice — Participants engaged in several different types of memory practice procedures on assigned laptops. The procedures focused on memory for action plans for screening and condom use.
  Arms: Memory Practice

SUMMARY:
A randomized trial was conducted at drug diversion educational programs with a sample of 343 adult drug offenders who volunteered for the study. The trial tested three different interventions on HIV testing and condom use, with a 3 month follow-up. The study translated consistent basic research showing strong effects of memory practice on memory for new material. One of the conditions involved extensive memory practice of action plans involving HIV testing and condom use. Other conditions varied two active control interventions. Results showed that the memory practice condition led to a substantially larger odds of HIV testing than did the two control conditions. Condom use was also significantly more frequent in the memory practice condition than in one of the control conditions but was not significantly different from the second control condition.

DETAILED DESCRIPTION:
This study translated basic research from several areas of cognitive science to a new intervention procedure designed to reduce HIV risk and increase screening for HIV and other infections. A randomized trial was conducted (N = 343) to test effects on testing for infection (HIV and hepatitis B/C) and condom use frequency in a sample of drug offenders at risk for infection. Many populations of drug offenders are not currently receiving evidence-based prevention for HIV or hepatitis and are in need of effective interventions that can be used in existing drug programs. At three-month follow-up, the results revealed that the condition translating basic research on memory practice and integrative processing significantly increased the odds of infection testing as compared to two alternative conditions. This condition also significantly improved the extent of condom use, compared to a traditional health education condition. The results show promise for increased translation of basic research on memory to behavioral interventions on health and prevention science. Such procedures can be effectively applied in a complex field setting in existing drug diversion programs.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in drug diversion education program
* Minimum age 18
* Understand English

Exclusion Criteria:

* Under 18
* Do not understand English
* Obviously intoxicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2013-10-15 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2016-03-31 (Actual)

PRIMARY OUTCOMES:
HIV and other infection testing | Past 3 months
  HIV testing was measured with items from the National Sexual Health Survey (Catania et al., 1992). Hepatitis testing items were assessed in an identical structure. Testing for other sexually transmitted diseases was measured with items from the AIDS Risk Behavior Assessment (Donenberg et al., 2001). These items were tabulated to form a binary variable of whether participants reported testing for HIV, hepatitis, or other sexually transmitted diseases within the past 3 months (3 months following intervention).
Condom use | Past 3 months
  Condom use was assessed with three condom use frequency items from the HIV Risk-taking Behavior Scale (Darke et al., 1991; α =.70; test-retest, r = .86). Response agreement between participants and their sex partners ranged from 88% to 100% in previous research. The questions asked how often participants used condoms in the past 3 months (following the intervention) when having vaginal, oral, or anal sex on a 5-point scale: never, some of the time, about half of the time, most of the time, always.

IPD SHARING:
Plan to Share IPD: Yes
Pretest and outcome data will be made available after publication. Data can be obtained from the PI at alan.stacy@cgu.edu

REFERENCES:
- [Background] Catania JA, Coates TJ, Stall R, Turner H, Peterson J, Hearst N, Dolcini MM, Hudes E, Gagnon J, Wiley J, et al. Prevalence of AIDS-related risk factors and condom use in the United States. Science. 1992 Nov 13;258(5085):1101-6. doi: 10.1126/science.1439818.
- [Background] Donenberg GR, Emerson E, Bryant FB, Wilson H, Weber-Shifrin E. Understanding AIDS-risk behavior among adolescents in psychiatric care: links to psychopathology and peer relationships. J Am Acad Child Adolesc Psychiatry. 2001 Jun;40(6):642-53. doi: 10.1097/00004583-200106000-00008. PMID 11392341
- [Background] Darke S, Hall W, Heather N, Ward J, Wodak A. The reliability and validity of a scale to measure HIV risk-taking behaviour among intravenous drug users. AIDS. 1991 Feb;5(2):181-5. doi: 10.1097/00002030-199102000-00008. PMID 2031690
- See also: website with HIV related videos used in intervention — http://aidsvideos.org/